CLINICAL TRIAL: NCT01726725
Title: Investigating the Etiology of Hemifacial Spasm (HFS): The Role of Desflurane
Brief Title: Hemifacial Spasm and Desflurane
Acronym: HFS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Other Study IDs: B2012:099
Record Dates: First submitted 2012-11-07; First posted 2012-11-15 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: Hemifacial Spasm
Keywords: hemifacial spasm; microvascular decompression surgery; desflurane
MeSH Terms: conditions — Hemifacial Spasm | interventions — Desflurane

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- hemifacial spasm, lateral spread, motor evoked potentials: EMG recordings from facial muscles of HFS patients during MVD surgery will be compared during total intravenous anesthesia (propofol), 0.5 MAC desflurane and 1.0 MAC desflurane
  Interventions: Drug: desflurane

INTERVENTIONS:
Drug: desflurane

SUMMARY:
Patients are chosen to participate in this study because they will undergo a particular type of brain surgery to treat their hemifacial spasm. This surgery is called microvascular decompression (MVD) and involves the facial nerve. The facial nerve is being compressed by one or more blood vessels and this contact produces the facial twitches. The investigators do not know why a blood vessel that touches the facial nerve produces facial twitches. The investigators are interested in investigating this during your surgery. A total of 25 participants are expected to participate in this study.

DETAILED DESCRIPTION:
"Intra Operative Monitoring" (IOM) is a standard and routine medical practice for patients having MVD surgery. IOM is done to make sure that the hearing and face nerves are not accidentally bumped or damaged during surgery. After anesthetic induction, the neurophysiologist places electrodes for the nerves, on the scalp and muscles. Stimulation and monitoring of muscle twitches are all common, safe and painless medical procedures.

In this study, the investigators would like to measure the nerve and muscle function on the normal side and compare it to nerve and muscle function on the abnormal side during different levels of the anesthetic desflurane. In order to monitor the normal side of the face one additional set of electrodes will be placed in the facial muscles. The investigators will compare responses to three different levels of anesthetic. The technique used will be motor evoked potentials. The effect of the anesthesia on the lateral spread response will also be examined. This response is evident only on the symptomatic side. These observations will take approximately 10 to 15 minutes and will not delay or lengthen the surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients referred to the neurosurgical service for microvascular decompression surgery for HFS
* males and females 18 to 75 years of age
* otherwise normal neurological exam
* signed informed consent

Exclusion Criteria:

* Botox treatment within the last three months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with hemifacial spasm who will be undergoing microvascular decompression surgery
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Measure EMG responses to peripheral nerve stimulation and motor cortex stimulation during changes in desflurane levels | one year

CONTACTS AND LOCATIONS:
Overall Officials: Marshall Wilkinson, PhD, Principal Investigator — University of Manitoba